CLINICAL TRIAL: NCT04589728
Title: Prospective and Retrospective Observational Evaluation of Real World Outcome of Unfit Patients With Acute Myeloid Leukemia Treated With the Combination Venetoclax Plus Hypomethylating Agents, Under the Italian Law No.648/96
Brief Title: Prospective and Retrospective Observational Evaluation of Real World Outcome of Unfit AML Patients Treated With the Combination Venetoclax Plus Hypomethylating Agents, Under the Italian Law No.648/96
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML2320
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: venetoclax; unfit AML patients; Hypomethylating agents
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients being observed during the study duration.
  Interventions: Drug: Venetoclax plus HMA

INTERVENTIONS:
Drug: Venetoclax plus HMA — patients with AML, ineligible for intensive chemotherapy, treated with the combination of HMA plus venetoclax under the Italian Law N. 648/96.

SUMMARY:
This is an retrospective and prospective observational multinstitutional study to evaluate the impact on outcome of the combination of HMA plus venetoclax in AML patients unfit for intensive chemotherapy in a "real-life" scenario. No additional procedures or visits other than those required by normal clinical practice will be required. Patients will be observed for at least 24 months.

DETAILED DESCRIPTION:
This is an retrospective and prospective observational multinstitutional study to evaluate the impact on outcome of the combination of HMA plus venetoclax in patients with AML unfit for intensive chemotherapy in a "real-life" scenario. At least 104 AML adult patients ineligible for intensive chemotherapy treated with the combination HMA plus venetoclax under the Italian Law No.648/96 by December 2021 will be enrolled. No additional procedures or visits other than those required by normal clinical practice will be required. Patients will be observed for at least 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with a diagnosis of previously untreated primary or secondary AML;
* Deemed ineligible for intensive chemotherapy because of age (≥75 years), performance status or comorbidities as defined by the treating physicians, according to SIE/SIES/GITMO criteria;
* Eligible to receive the combination HMA plus venetoclax under the Italian Law No.648/96 by December 2021;
* Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* Acute promyelocytic Leukemia;
* Previous first-line treatments for AML;
* Previous treatments with HMA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of AML ineligible for intensive chemotherapy treated with the combination HMA plus venetoclax under the Italian Law No.648/96 by December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 15 months
  Evaluation of Overall Survival in AML patients ineligible for intensive chemotherapy treated with the combination of HMA plus Venetoclax

CONTACTS AND LOCATIONS:
Locations (23):
- Italy (23):
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Aou Ospedali Riuniti - Foggia - Uoc Ematologia, Foggia
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Istituto Europeo Di Oncologia Irccs - Milano - Divisione Di Oncoematologia, Milan
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Ao Regionale S. Carlo - Potenza - Sic Ematologia, Potenza
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari
  - Ospedale Di Sassuolo Spa - Ematologia, Sassuolo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Asl Di Viterbo, Complesso Ospedaliero Di Belcolle - Uoc Ematologia, Viterbo